CLINICAL TRIAL: NCT05936346
Title: Evaluation of Safety and Tolerability of Salvia Haenkei Extract As a Dietary Supplement Ingredient in a Healthy Population: a Randomized, Open Label, Parallel-arm, Two-dose Study
Brief Title: Evaluation of Safety and Tolerability of Salvia Haenkei Extract As a Dietary Supplement Ingredient
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IBSA Farmaceutici Italia Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB-IT-SAL-22
Record Dates: First submitted 2023-06-22; First posted 2023-07-07 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Aging

STUDY DESIGN:
Intervention Model Description: Randomized, Open label, Parallel-arm, Two-dose Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lower dose (175mg) (Experimental): The study intervention consists of a single daily oral intake 175 mg of Salvia haenkei as soft capsule over a period of 3 months.
  Interventions: Dietary Supplement: Salvia haenkei 175mg
- Higher dose (350mg) (Experimental): The study intervention consists of a single daily oral intake 350 mg of Salvia haenkei as soft capsule over a period of 3 months.
  Interventions: Dietary Supplement: Salvia haenkei 350mg

INTERVENTIONS:
Dietary Supplement: Salvia haenkei 175mg — The product appears as a soft gel containing the dry extract of Salvia haenkei
  Arms: Lower dose (175mg)
Dietary Supplement: Salvia haenkei 350mg — The product appears as a soft gel containing the dry extract of Salvia haenkei
  Arms: Higher dose (350mg)

SUMMARY:
Evalution of the safety and tolerability of the oral administration of Salvia haenkei in a healthy population.

DETAILED DESCRIPTION:
The aim of the study is to assess the safety and tolerability of the oral administration of Salvia haenkei in a healthy population. Furthermore, Salvia haenkei has been identified as a potential anti-senescence agent and may counteract aging and aging-associated disorders. In this scenario, the current study aims also at exploring the effects of this supplementation on muscular and other organ functions (kidney, liver, heart, etc.) and on systemic inflammation and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Male or female
* Age 55-65 years, inclusive
* In good general health as evidenced by medical history and current health status
* Willingness to maintain dietary and sports habits as of baseline
* Willingness and ability to comply with the requirements of the study

Exclusion Criteria:

* Body Mass Index < 18.5 or ≥ 30
* Difficulty in swallowing (dysphagia)
* Known allergy or sensitivity to any ingredient of the study intervention
* Any medical condition or clinically significant abnormalities in laboratory values (hematology, blood chemistry, urinalysis) at screening which in the judgment of the Investigator makes the subject unsuitable for the study
* Planned or anticipated major surgical procedure during the subject's participation in this study
* Inability or contraindications to undergo the study intervention
* Inability to follow the procedures of the study (e.g. due to language problems, psychological disorders, dementia, etc.)
* Use of any new vitamins, herbal or dietary supplements, functional foods and sports drink, of any kind, liable or presented as liable to enhance physical performances within one month prior to the start and during the study

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events | From Day 0 to Day 90
  Number of adverse events, serious adverse events, clinically significant changes in clinical laboratory assessments (hematology, chemistry, urinalysis) and clinically significant changes in vital signs or other clinical assessments will be evaluated.
Tolerability assessment by evaluation of the number of subjects who will not withdraw prematurely from the study | From Day 0 to Day 90
  Tolerability is defined as the number of subjects who will not withdraw prematurely from the study due to the occurrence of any AEs or SAEs.

SECONDARY OUTCOMES:
Change from baseline of muscle strength assessed by grip test using the pneumatic dynamometer | Day 0, Day 90
  Subjects will be asked to squeeze rubber balls (available in three sizes) three times for each side using the dominant hand. The best result of the 3 attempts will be taken into consideration.
Change from baseline of muscle strength assessed by repeated chair stand test | Day 0, Day 90
  Repeated chair stand test is a timed test requiring subjects to rise from a chair without using their arms and return to the seated position, consecutively, for five times. This test has been shown to be able to provide a reliable and valid indication of lower body strength. The cut-off is > 15 seconds for five rises.
Change from baseline of physical performance assessed by gait speed test | Day 0, Day 90
  Gait speed test is used to assess walking speed in meters per second over a 4-metre distance at a comfortable pace. Subjects with a gait speed <0.8 m/s are described as having a poor physical performance.
Change from baseline of physical performance assessed by six minute walking test | Day 0, Day 90
  The six minute walking test will assess functional exercise capacity. The test will measure the distance that a subject can quickly walk on a flat, hard surface in a period of 6 minutes. It evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units, and muscle metabolism.
Change from baseline of muscle mass assessed by BMI calculation (weight/height^2) | Day 0, Day 90
  Muscle mass will be measured BMI calculation (weight/height^2)
Change from baseline of muscle mass assessed by calf circumference measurement (cm) | Day 0, Day 90
  Muscle mass will be measured using calf circumference (maximum circumference of calf of lower non-dominant leg bent at 90 degrees, cut-off <31 cm)
Change from baseline of muscle mass assessed by mid-upper arm circumference measurement (cm) | Day 0, Day 90
  Muscle mass will be measured using mid-upper arm circumference (circumference at halfway point between the olecranon process and acromion while arm is bent at 90 degrees, cut-off <22.5 cm).
Change from baseline of the risk of sarcopenia assessed by SARC-F questionnaire | Day 0, Day 90
  The subject will be asked 5 questions addressing strength, assistance in walking, rising from a chair, stair climbing and falls. Each component is scored from 0 to 2 points, giving a global score of the SARC-F between 0 and 10 points. A score ≥ 4 points is reported to be predictive of sarcopenia and poor outcomes.
Change from baseline of muscle echogenicity assessed by muscle ultrasound | Day 0, Day 90
  Muscle echogenicity will be measured using a semi-quantitative scale
Change from baseline of muscle thickness assessed by muscle ultrasound | Day 0, Day 90
  Muscle thickness (mm) will be measured by muscle ultrasound
Change from baseline of DNA Methylation | Day 0, Day 90
  Assessment of methylation status in 353 CpG sites associated with aging from DNA in whole blood. The analysis of DNA Methylation will be done only for the 25 subjects enrolled to the high dosage arm [350 mg]) (translational endpoint)
Change from baseline of the amount of blood biomarkers indicative of aging, metabolism and inflammation | Day 0, Day 45, Day 90
  Blood biomarkers indicative of aging, metabolism and inflammation including cytokines and other relevant biomarkers will be quantified by ELISA (translational endpoint)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Noseda, MD, PhD, Principal Investigator — Istituto di Scienze Farmacologiche della Svizzera Italiana, Lugano (Switzerland)
Locations (1):
- Ospedale Regionale di Lugano, Lugano, Switzerland